CLINICAL TRIAL: NCT04242225
Title: Accuracy of Using 2D Transesophageal Echocardiography Compared to Balloon Sizing in Determining Valve Size During Transcatheter Aortic Valve Implantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Collaborators: Duisburg Heart center ,Dusseldorf University ,Germany (Unknown)
Responsible Party: Principal Investigator, Marwan Sayed Mahmoud, Assiut university Heart Hospital, Assiut University
Other Study IDs: AssiutUni
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Aortic Stenosis, Calcific
MeSH Terms: conditions — Aortic Valve, Calcification of

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The method of transcatheter aortic valve implantation (TAVI) introduced in 2002 by Alain Cribier et al. has offered new prospects for patients with severe aortic stenosis and multiple comorbidities, who are at high operative risk(1).

The PARTNER series of randomized controlled trials has firmly established the role of TAVI with the balloon-expandable Edwards Sapien valve in patients with severe symptomatic aortic stenosis (AS) at prohibitive risk of surgery (PARTNER IA), high risk for surgery (PARTNER IB), and intermediate risk for surgery (PARTNER 2).(2)

Also PARTNER 3 and Evolut Low Risk trial strongly suggest that TAVI is not only a suitable alternative and may be superior to surgical aortic valve replacement ( SAVR) in low-risk patients.(2)

The accurate determination of the size of the implant is dependent on pre-procedural imaging. Annular measurements are important in the TAVI as inaccurate estimation can lead to complications e.g paravalvular leakage .(3) Transthoracic echocardiography (TTE), transoesophageal echocardiography (TOE), multidetector computed tomography (MDCT) and magnetic resonance imaging (MRI) have been extensively studied with respect to pre-procedural aortic annular sizing.(3).

However, even with some of the evidence returning a discrepancy in annular measurements between techniques, the literature to date does not clarify whether TOE undersizes inappropriately or appropriately with respect to MDCT.(3) In a recent study, 29.5% of patients would have been deemed ineligible for TAVI because of overestimation of annular measurements by MDCT, a figure reduced to 1.3% with the use of TOE (4)

In a recent small retrospective study, TOE, MDCT and MRI all performed comparatively well with device sizing. (5)

Balloon aortic valvuloplasty (BAV) dilatation before TAVI is considered a mandatory procedural step in the early years of TAVR. BAV is used to confirm annular sizing and to enhance trans-catheter heart valve (THV) deliverability.(6) However till now there is no comparison of annular measurement by 2D transesophgeal echocardiography with balloon sizing.

DETAILED DESCRIPTION:
Aim of work To compare accuracy of 2D transesophageal echocardiography versus balloon sizing in determining size of device during transcatheter aortic valve implantation and inhospital outcomes of this approach using 2D TEE and balloon sizing only during TAVI .

Patients and methods. The study will include (100) patients, prospective observational study

All patient will undergo :

1-Written consent. 2-Detailed history including symptoms (NYHA class) ,co morbidities 3-Clinical examination 4-Electrocardiogram (detection of conduction disturbance , ischemic changes). 5-Laboratory investigation (hemoglobin level, creatinine, glomerular filteration rate(GFR)) 6-Risk stratification: using STS score 6- Transthoracic Echocardiography: (7)

1-Assesment of aortic valve by

1. Mean and maximum pressure gradiant (severe AS if mean pressure >40mmhg and maximum pressure >64mmhg) in presence of normal ejection fraction (EF).
2. Aortic valve area by continuity equation (severe AS if < 1cm2).
3. Measurement of aortic valve annulus (in parasternal long axis view) .
4. Assesment of associated aortic regurge (8) :

   -Regurge jet width/LVOT width (mild <25%,moderate 25-65%, severe >65%)
   * Vena contracta (VC) (mild <0.3cm, moderate 0.3-0.6cm, severe >0.6cm)
   * Regurge volume (RV) (mild <30ml, moderate 30-60ml, severe >60ml).
   * Regurge fraction (RF) (mild <30%, moderate 30-50% and severe > 50%).
   * Effective regurgitant orifice area (EROA) (mild <0.1 cm, moderate 0.1-0.29cm and severe ≥0.3cm) 2- Assesment of EF (by M-mode and simpsons method). 3-Assesment of other valves .

     7-Transesophegeal Echocardiography.(9):
     1. Morphology of valve (tricuspid, bicuspid , unicuspid).
     2. Measurement of aortic valve area (AVA) by planimetry.
     3. Extent, distribution and location of Calcification. (annular calcification symmetrical or asymmetrical, sinuotubular junction , subvalvular calcification)
     4. Measurement of aortic annulus dimension, LVOT, sinus of valsalva, sinotubular junction and ascending aorta dimensions.

   Determinations of 2D TEE aortic annular and LVOT diameters were performed in the 3-chamber long-axis view at approximately the 120◦ angle during early systole . The aortic annular diameter was measured from the junction of the aortic leaflet with the septal endocardium to the junction of the leaflet with the mitral valve posteriorly, using the inner edge to inner edge. The LVOT diameter was obtained 5 mm into the LVOT from the level of the annulus.(10) Calculation of a cover index: defined as a 100 x (prosthesis diameter - transoesophageal echocardiography annulus diameter)/prosthesis diameter. (11).

   6- Aortic atheroma: The Katz classification for grading aortic atheromas is as follows: Grade 1, normal-appearing intima of the aorta; Grade 2, extensive intimal thickening; Grade 3, sessile atheroma protruding <5 mm into the aorta; Grade 4, sessile atheroma protruding >5 mm; and Grade 5, mobile atheroma.(12) 7-Associated basal septal hypertrophy . 8-Assesment of associated aortic regurge. 8-Pre-TAVI workup in cardiac catheterization laboratory:
   1. Access route evaluation: assess peripheral vasculature for size, tortuosity, calcification -Iliofemoral angiography: A 5F metric (graded) pigtail is used for calibration and accurate determination of vessel calibre and minimal lumen diameter. The pigtail is placed at the lumber 4/5 level, which approximates a position just proximal to the common iliac bifurcation with injection of 15-20mls contrast at 20mls/sec.

      -Iliofemoral diameter: determined by Sheath-to-iliofemoral artery ratio (SIFAR) was defined as sheath outer diameter divided by access-side vasculature diameter.

      -Iliofemoral calcification: Calcification can be evaluated on fluoroscopy and graded as: none, mild (spotty), moderate (coalescing), severe (bulky, protruding, horse-shoe, circumferential ). Iliofemoral tortuosity : determined by tortuosity score which is defined as follows: 0 = no tortuosity; 1 = mild tortuosity (30° to 60°); 2 = moderate tortuosity (60° to 90°); and 3 = marked tortuosity (>90°).(13)

      -Subclavian or axillary angiography if femoral axis is unsuitable.
   2. Diagnostic coronary angiography: for assessment of presence and severity of coronary artery disease.
   3. Aortogram: is done to asses for angle between LVOT and ascending aorta , distance of coronary vessels from annulus and presence of aortic regurge.

      * 5F graded pigtail is placed into the non-coronary cusp (NCC) and an aortogram performed (20mls contrast at 20mls/sec). Fluoroscopic projection of RAO 30◦ and LAO 30◦.
   4. Aortic valve cross over: to demonstrate feasibility of crossing valve.
   5. Hemodynamic assessment: assess invasive transaortic gradiant with simultaneous pressure transduction.

      * Pigtail will be crossed into the LV cavity, simultaneous measurement of pressures from the LV and femoral artery can be obtained. Use of a 5F pigtail enables simultaneous pressures to be transduced from the 6F femoral artery sheath without the need for a second arterial sheath.
   6. Left ventriculogram: assess EF by eyeballing (mild 40-50%,moderate 30-40% and severe <30%) and presence of MR according to seller criteria described later on.

      Left ventriculography is done using 25ml contrast at rate 10ml/second in both RAO 30◦ and LAO 60◦
   7. Right heart catheterization: assess pulmonary artery (PA) pressure, Pulmonary capillary wedge pressure (PCWP).

   TAVI procedure:

   The detailed steps of procedure are reported by Nijhoff F,etal. TAVI is performed through transfemoral or transapical approach, based on the feasibility of the iliofemoral anatomy and suitable access sites. All procedures are performed in a fully equipped hybrid cardiac catheterization laboratory. Surgical cutdown is used to close the vascular access site at the femoral arteries.

   Fluoroscopy is used to guide the deployment of the valves and prosthesis positioning. Both predilatation of the native valve and prosthetic valve implantation are performed during rapid right ventricular pacing (160 to 200 beats/min). Prosthesis position, function, and coronary ostia patency are assessed with fluoroscopy and aortography .

   -Balloon sizing: An appropriately sized valvuloplasty balloon is choiced .The initial volume of inflation is set to obtain a balloon size of 1 mm less than the TEE measurement. The balloon is positioned across the aortic valve through femoral sheath and inflated with the same volume during rapid ventricular pacing, using a 30 cc inflation syringe.

   At full inflation, an aortography is performed. The following parameters are recorded: (I) presence of a waist on the balloon at the level of the annulus, (II) intra-balloon pressure, (III) patency of the coronary artery ostia and their relations with the displaced aortic valve cusps, (IV) presence and entity of aortic regurgitation on aortography at full balloon inflation ("para-balloon leak"). In the absence of a waist on the balloon and/or in case of major para-balloon leak, the procedure is repeated with a larger diameter balloon (larger balloon or same balloon inflated with a larger volume of contrast media).

   Assesment of inhospital outcomes after TAVI procedure:

   1- paravalvular leakage : Assessment of paravalvular leakage

   1-Angiographic evaluation of paravalvular leakage :

   Ten minutes after the deployment of the prosthetic valve, angiography of the aortic root is performed to assess the severity of aortic regurgitation according to Sellers criteria (14):

   (0) no regurgitation.
   1. only trace of contrast could be seen in the left ventricle, and it is cleared in each systole.
   2. contrast filling the entire LV in diastole with less density compared with opacification of the ascending aorta.
   3. contrast filling the entire LV in diastole equal in density to the contrast opacification of the ascending aorta.
   4. contrast filling of the entire LV in diastole on the first beat with greater density compared with the contrast opacification of the ascending aorta.

   Two observers independently score the images. In case of discrepancy the images will be re-evaluated and consensus will be reached by a third observer. .

   2-Transthoracic Echocardiographic study:

   All patients will be evaluated after TAVI by pre-discharge transthoracic echocardiography. The extent of PVL is assessed according to the main VARC criteria (15):

<!-- -->

1. Semiquantitative parameters

   1. Diastolic flow reversal in the descending aorta-pulsed wave : mild (Absent or brief) ,moderate ( early diastolic Intermediate), severe (Prominent holodiastolic)
   2. Circumferential extent of prosthetic valve paravalvular regurgitation:

   (0) no regurgitation; (1) mild PVL is defined as<10 % circumferential extent; (2) moderate PVL was defined as [>10 % but<30 % of PVL and (3) severe PVL is defined as >30 % according to the updated VARC guideline , that is the circumferential extent of PVL in a parasternal short-axis view (19).
2. Quantitative parameters:

   1. Regurgitant volume (ml/beat) mild (<30) , moderate (30-59) ,severe (>60).
   2. Regurgitant fraction (%) mild (< 30), moderate (30-49 ) ,severe (>50).
   3. Effective regurgitant orifice area (cm2) mild (<0.10) ,moderate (0.10-0.29) , severe (>0.30).

   2-Other complication results from inaccurate annular sizing : prosthesis embolization, annular rupture, aortic dissection, coronary artery occlusion , conduction defects.

   3-Assesment of other complication ,vascular site complication, bleeding, stroke and mortality.

   Statistical analysis:

   The collected data will be tabulated and statistically analyzed and will be shown in tables and figures.

ELIGIBILITY:
Inclusion Criteria:

* 1-Patients must have severe degenerative high flow AS (echocardiographic criteria: aortic valve (AV) effective orifice area (EOA) of < 1 cm2, mean AV gradient of > 40 mmHg, or AV peak systolic velocity of > 4.0 m/s) in presence of normal ejection fraction (EF).

  2- Patients must be symptomatic from the AS (dyspnea in NYHA-class II or greater, angina pectoris, or syncope), or asymptomatic but with decreased left ventricular ejection fraction, positive stress test , Pulmonary hypertension (systolic pulmonary artery pressure >60 mmHg).

  4-Symptomatic patients with severe low-flow, low-gradient (<40 mmHg) aortic stenosis with reduced ejection fraction and evidence of flow (contractile) reserve.

  3- Patients surviveal time more than one year . 4- Patients have contraindications for open chest surgery, such as :
  1. Presence of comorbidities not adequately reflected by risk scores.
  2. Procelain aorta
  3. Squelae of chest radiation.
  4. Severe chest deformation or scoliosis.
  5. Previous cardiac surgery

     Exclusion Criteria:
     1. Evidence of an acute myocardial infarction 30 days before the intended treatment.
     2. Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is noncalcified.
     3. Mixed aortic stenosis and aortic regurgitation with predominant aortic regurgitation > 3+).
     4. Hemodynamic or respiratory instability within 30 days of screening evaluation.
     5. Need for emergency surgery for any reason.
     6. Hypertrophic cardiomyopathy with or without obstruction.
     7. Severe left ventricular dysfunction with LVEF <20%.
     8. Severe pulmonary hypertension and RV dysfunction.
     9. Echocardiographic evidence of intracardiac mass, thrombus or vegetation. . 10-A known contraindication to all anticoagulation regimens, or inability to be anticoagulated for the study procedure.

     11-MRI confirmed stroke or transient ischemic attack within 6 months (180 days) of the procedure.

     12-Renal insufficiency (creatinine >3mg) and / or end stage renal insufficiency requiring chronic dialysis at the time of screening.

     13-Estimated life expectancy<12 month.

     . 14-Severe incapacitating dementia 15-Significant aortic disease, including abdominal aortic or thoracic aneurysm defined as maximal luminal diameter 5 cm or greater; marked tortuosity (hyperacute bend), aortic arch atheroma [especially if thick (>5 mm), protruding or ulcerated] or narrowing of the abdominal or thoracic aorta, severe tortuosity of the thoracic aorta.

     Also a minimum iliac or femoral artery diameter of less than 6 mm may be deemed unsuitable for femoral approach.

     16-Severe mitral regurgitation. 17-Annulus size out of range of available prosthese (<18mm and >29mm). 18-Untreated coronary artery disease requiring revascularization. 19- Elevated risk of coronary ostium obstruction (asymmetric valve calcification, short distance between annulus and coronary ostium less than 10mm.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with severe aortic stenosis presented for TAVI
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of 2D transesophgeal echocardiography compared to balloon sizining in determining size of valve during TAVI | 6 months
  accuracy of 2D transesophgeal echocardiography compared to balloon sizining in determining size of valve during TAVI

SECONDARY OUTCOMES:
in hospital outcomes of this approach using 2D TEE and balloon sizing only during TAVI | 6 months
  paravalvular leakage,conduction defects ,valve embolization ,...

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Sa Mahmoud, Master, Principal Investigator — Assiut University; Marwan Sa Mahmoud, Master, Principal Investigator — HZD
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No